CLINICAL TRIAL: NCT02835235
Title: A Double-blinded Placebo-controlled Multiple Dose Trial Investigating Safety, Tolerability, PK and PD for Multiple Doses of NNC9204-0530 in Male and Female Subjects Being Overweight or With Obesity
Brief Title: A Trial Investigating Safety, Tolerability, PK and PD for Multiple Doses of NNC9204-0530 in Male and Female Subjects Being Overweight or With Obesity
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: NN9030-4295; U1111-1180-3542 (Other: WHO)
Record Dates: First submitted 2016-07-13; First posted 2016-07-18 (Estimated); Last update posted 2018-01-08 (Actual); Status verified 2018-01

CONDITIONS: Metabolism and Nutrition Disorder; Obesity
MeSH Terms: conditions — Nutrition Disorders; Obesity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- NNC9204-0530 (Experimental): Dose-escalation within the cohort before reaching final dose
  Interventions: Drug: NNC9204-0530
- Placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: NNC9204-0530 — Administered daily subcutaneously (s.c., under the skin)
  Arms: NNC9204-0530
Drug: placebo — Administered daily subcutaneously (s.c., under the skin)
  Arms: Placebo

SUMMARY:
This trial is conducted in the United States of America. The aim of the trial is to investigate Safety, Tolerability, PK and PD for Multiple Doses of NNC9204-0530 in Male and Female Subjects being overweight or with obesity

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age between 18 and 55 years (both inclusive) at the time of signing informed consent
* Body mass index between 25.0 and 39.9 kg/m^2 (both inclusive) at screening.

Exclusion Criteria:

* Haemoglobin A1c (HbA1c) equal or above 6.5%
* Any clinically significant weight change (above or equal to 5% self-reported change) or dieting attempts (e.g. participation in an organized weight reduction program) within the last 90 days prior to screening
* Any prior obesity surgery or currently present gastrointestinal implant.
* Abnormal ECG (electrocardiogram) results including 2nd or 3rd degree AV-block, prolongation of the QRS complex above 120 ms, or the QTcF interval above 430 ms (males) or above 450 ms (females), or other clinically relevant abnormal results, as judged by the investigator
* A history of additional risk factors for Torsades de pointes (e.g., heart failure, hypokalaemia, family history of Long QT Syndrome)
* History of pancreatitis (acute or chronic)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2016-07-26 (Actual); Primary Completion 2017-07-07 (Actual); Study Completion 2017-07-07 (Actual)

PRIMARY OUTCOMES:
Number of treatment emergent adverse events | Day 1-112

SECONDARY OUTCOMES:
Area under the NNC9204-0530 serum concentration-time curve | Day 84-112
Time to maximum serum concentration of NNC9204-0530 | Day 84-112
Change in HbA1c | Day -1, Day 85

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (2):
- United States (2):
  - Novo Nordisk Investigational Site, Tempe, Arizona
  - Novo Nordisk Investigational Site, Lincoln, Nebraska

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com